



Title A Randomized, Placebo-controlled, Double-blind, Multicenter

Phase 2 Study of Atezolizumab With or Without Entinostat in Patients with Advanced Triple Negative Breast Cancer, with a

Phase 1b Lead in Phase

Study Number SNDX-275-0602 (TRIO025)

**Document Number** DM-025-037

Version Number 1.0

**Product Name** Entinostat (SNDX-275)

**Indication** Advanced Triple Negative Breast Cancer (aTNBC)

Study Phase 1b/2

**Sponsor** Syndax Pharmaceuticals, Inc.

400 Totten Pond Road, Suite 110

Waltham, MA 02154

Version Date 08-Jun-2017

#### **Confidentiality Statement**

The information contained herein is confidential and proprietary and may not be disclosed, reproduced, or circulated without the prior written consent of TRIO.

Document owner(s):


Document ID: DM-025-037 Version: 1.0 – Final – 08-Jun-2017

| STAT | TISTICAL ANALYSI | S PLAN APPROVAL | SHEET |
|---|---|---|---|
| Protocol Number: | SNDX-275-0602 (TR | IO025) <b>Product:</b> | Entinostat (SNDX-275) |
| Protocol Title: | | | |
| A Randomized, Placebo | -controlled, Double-bl | ind, Multicenter Phase | 2 Study of Atezolizumab |
| With or Without Entine | ostat in Patients with | Advanced Triple Nega | tive Breast Cancer, with a |
| Phase 1b Lead in Phase. | | | |
| Author: | | | |
| Version Number: | 1.0 | <b>Version Date:</b> | 08-Jun-2017 |
| The undersigned have re | viewed this plan and fi | nd it to be consistent w | ith the requirements of the |
| protocol as it applies to t | heir respective areas. | | |
| | | Date | Signature |
| | , TRIO | | |
| , TI | RIO | | |
| , TRIO | | | |
| , T | RIO | | |
| , 7 | ΓRIO | | |

| STATISTICAL | ANALYSI | S PLAN APPROVAL | SHEET |
|---|---|---|---|
| SNDX-275-0602 (TRIO025) | <b>Product:</b> | Entinostat (SNDX-27: | 5) |
| Protocol Title: | | | |
| A Randomized, Placebo-controlled, | Double-blin | d, Multicenter Phase 2 | Study of Atezolizumab With |
| or Without Entinostat in Patients w | ith Advance | ed Triple Negative Bre | ast Cancer, with a Phase 1b |
| Lead in Phase. | | | |
| Author: | | | |
| Version Number: 1.0 | | Version Date: | 08-Jun-2017 |
| The undersigned have reviewed this | plan and fi | nd it to be consistent i | with the requirements of the |
| protocol as it applies to their respect | ive areas. | | |
| | | Date | Signature |
| Scott Cruickshank & Associates | | | |
| | , | | |
| Syndax Pharmaceuticals, Inc. | | | |
| Syndax Pharmacueticals, Inc. | | | |

# TABLE OF CONTENTS

| | Introduction | |
|----|--------------------------------------------------------------------|----|
| 2. | Study Objectives | 10 |
| | 2.1 Primary Objective | 10 |
| | 2.2 Secondary Objectives | 10 |
| | 2.2.1 Efficacy | |
| | 2.2.2 Safety | |
| | 2.3 Exploratory Objectives | |
| 3. | Study Design | |
| ٠. | 3.1 Phase 1b Dose Determination Phase | |
| | 3.2 Phase 2 Expansion Phase | |
| 4 | Study Endpoints | |
| ٠. | 4.1 Phase 1b Dose Determination Phase | |
| | 4.2 Phase 2 Expansion Phase | |
| | 4.2.1 Primary Efficacy Endpoint | |
| | 4.2.2 Secondary Efficacy Endpoints | |
| | 4.2.3 Safety | |
| | 4.2.4 Exploratory | |
| 5. | <u>. </u> | |
| ٥. | 5.1 Hypothesis for Phase 2 | |
| | 5.2 Sample Size | |
| | 5.2.1 Phase 1b Dose Determination Phase | |
| | 5.2.2 Phase 2 Expansion Phase | |
| | 5.2.2 Phase 2 Expansion Phase 5.3 Randomization and Stratification | |
| | 5.4 Timing of Analyses | |
| | 5.4.1 Phase 1b Dose Determination Phase | |
| _ | 5.4.2 Phase 2 Expansion Phase | |
| 6. | Definitions | |
| | 6.1 Progression-Free Survival (PFS) | |
| | 6.2 Objective Response Rate (ORR) | |
| | 6.3 Clinical Benefit Rate (CBR) | |
| | 6.4 Overall Survival (OS) | |
| | 6.5 Duration of Response (DOR) | |
| | 6.6 Time to Response (TTR) | |
| | 6.7 Dose-limiting Toxicity (DLT) | |
| | 6.8 Maximum Tolerated Dose (MTD) | |
| | 6.9 Recommended Phase 2 Dose (RP2D) | |
| | 6.10 Treatment Emergent Adverse Events (TEAEs) | |
| | 6.11 Other Definitions | |
| | 6.11.1 Baseline | |
| | 6.11.2 Date of First Dose | |
| | 6.11.3 Date of Last Dose | |
| | 6.11.4 Last Contact Date | |
| 7. | | |
| | 7.1 Full Analysis Set (FAS) | |
| | 7.2 Per-protocol Analysis Set | 23 |


| | 7.3 | Safety Analysis Set | 23 |
|----|----------|-----------------------------------------------------|----|
| 8. | Inter | rim Analysis and Early Stopping Rule | 23 |
| 9. | Data | Screening and Acceptance | 23 |
| | 9.1 | General Principles | 24 |
| | 9.2 | Unblinding Plan | 24 |
| | 9.3 | Data Handling and Electronic Data Transfer. | 24 |
| | 9.4 | Handling of Incomplete and Missing Data | 25 |
| | 9.5 | Outliers | |
| | 9.6 | Validation Plan | 26 |
| 10 | ). Stati | stical Methods of Analysis | 26 |
| | 10.1 | Patient Disposition | 26 |
| | 10.2 | Demographics and Disease Characteristics | 27 |
| | 10.3 | Prior Surgery for Breast Cancer | 28 |
| | 10.4 | Prior Systemic Anti-Cancer Therapy | 28 |
| | 10.5 | Prior Radiation Therapy | 28 |
| | 10.6 | Medical History | 28 |
| | 10.7 | Extent of Exposure | 28 |
| | 10.8 | Efficacy Analyses | |
| | 10. | 8.1 PFS | 29 |
| | 10. | 8.2 ORR | 31 |
| | 10. | 8.3 CBR | 31 |
| | | 8.4 OS | |
| | 10. | 8.5 DOR and TTR | 31 |
| | 10. | 8.6 Anticancer therapy after end of study treatment | 31 |
| | 10.9 | | |
| | 10. | 9.1 Physical Examinations | 32 |
| | 10. | 9.2 Adverse Events | 32 |
| | | 9.3 Death | |
| | 10. | 9.4 Laboratory Values | 33 |
| | | 9.5 ECOG Performance Status | |
| | 10. | 9.6 Vital Signs | 33 |
| | | 9.7 Electrocardiogram (ECG) | |
| | | 9.8 Concomitant Medication | |
| | | Subgroup Analysis | |
| | | Pharmacokinetic and Antidrug Antibody Analyses. | |
| | | Correlative Analyses | |
| 11 | . List | of Planned Tables, Figures, Listings | |
| | 11.1 | Planned Tables | |
| | 11.2 | Planned Listings | |
| | 11.3 | Planned Figures | 42 |

#### **List of Abbreviations**

ADaM Analysis Data Model

ADSL Subject-level Analysis Dataset

AEs Adverse Events

aTNBC Advanced Triple Negative Breast Cancer

CBR Clinical Benefit Rate

CI Confidence Interval

CMH Cochran-Mantel-Haenszel

CR Complete Response

CTCAE Common Terminology Criteria for Adverse Events

DLT Dose-limiting Toxicity

DOR Duration of Response

DSMB Data Safety Monitoring Board

ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF electronic Case Report Form

FAS Full Analysis Set

FASFL Full Analysis Set Population Flag

HER2 Human Epidermal Growth Factor Receptor 2

irRECIST Immune-related RECIST

IDDI International Drug Development Institute

IV Intravenous

IWRS Interactive Web Response System

KM Kaplan-Meier

MedDRA Medical Dictionary for Regulatory Activities

MTD Maximum Tolerated Dose

NCI National Cancer Institute

NE Not evaluable

ORR Objective Response Rate

OS Overall Survival

PD Progressive Disease

PFS Progression Free Survival

PO per os (Oral Administration)

PPROTFL Per-protocol Population Flag

PR Partial Response

PT Preferred Term

Q1 First Quartile (25<sup>th</sup> percentile)

O3 Third Quartile (75<sup>th</sup> percentile)

RDI Relative Dose Intensity

RECIST Response Evaluation Criteria in Solid Tumors

RP2D Recommended Phase 2 Dose

SAEs Serious Adverse Events

SAFFL Safety Population Flag

SAP Statistical Analysis Plan

SD Stable Disease

SOC System Organ Class

Treatment Emergent Adverse Events **TEAEs** 

Tables, Listings, and Figures TLF

Translational Research in Oncology **TRIO** 

Time To Response TTR

World Health Organization Drug Dictionary WHODD

# **Revision History**

Not applicable; this is the initial version of Statistical Analysis Plan.

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes the detailed statistical methodology for executing the statistical analyses to assess the antitumor activity and safety profile of atezolizumab in combination with entinostat versus atezolizumab alone in treatment of advanced triple negative breast cancer (aTNBC) according to SNDX-275-0602 (TRIO025) protocol version 1.0.

Statistical analysis will be performed by TRIO using SAS® software Version 9.3 which meets the requirement as stated in the protocol.

#### 2. STUDY OBJECTIVES

# 2.1 Primary Objective

The primary objective for each phase of the study is as follows:

<u>Phase 1b (Dose Determination Cohort)</u>: To determine the dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of entinostat (SNDX-275) given in combination with atezolizumab.

<u>Phase 2 (Expansion Cohort):</u> To perform an evaluation of the efficacy of entinostat at the RP2D in combination with atezolizumab in patients with aTNBC, as determined by the duration of progression-free survival (PFS) based on the local investigator's assessment of progressive disease Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

# 2.2 Secondary Objectives

#### 2.2.1 Efficacy

To evaluate the efficacy of entinostat in combination with atezolizumab in patients with aTNBC, as determined by:

- PFS based on immune-related RECIST (irRECIST)
- Overall response rate (ORR) (complete response [CR] or partial response [PR]) based on RECIST 1.1
- ORR (irCR or irPR) based on irRECIST
- Clinical benefit rate (CBR) (CR or PR or stable disease [SD] for at least 24 weeks) based on RECIST 1.1
- CBR (irCR, irPR or irSD for at least 24 weeks) based on irRECIST
- Overall survival (OS)

In patients with best overall response of CR or PR based on RECIST 1.1 and irCR or irPR based on irRECIST:

- Duration of response (DOR)
- Time to response (TTR)

# 2.2.2 Safety

To evaluate safety and the tolerability of entinostat in combination with atezolizumab, as measured by clinical adverse events (AEs) and laboratory parameters.

# 2.3 Exploratory Objectives

The exploratory study objectives are to:

| • | |
|---|---|
| | · |
| • | |
| • | |
| _ | |
| • | |
| • | |
| • | |
| • | |
| • | |
| • | |
| • | |
| • | |
| • | |

The exploratory objectives will be performed afterwards and detailed in a separate document(s).

# 3. STUDY DESIGN

This is a Phase 1b/2 study evaluating the combination of entinostat plus atezolizumab in patients

with aTNBC. The study has 2 phases: an open-label Dose Determination Phase (Phase 1b) followed

by an Expansion Phase (Phase 2).

The Expansion Phase will evaluate the efficacy and safety of entinostat when administered at the

RP2D with atezolizumab in patients with aTNBC in a randomized, double-blind, placebo-

controlled setting.

3.1 Phase 1b Dose Determination Phase

This study phase employs a classical 3+3 design, with the determination of DLT and the MTD or

RP2D at cycle 1 based on the combination of entinostat (at the dose of 5mg, 3mg or 2mg weekly)

with atezolizumab at a fixed dose of 1200 mg iv. Six patients will need to be treated in a dose level

for it to be considered MTD or the RP2D. The recommended dose for Phase 2 investigation will be

the higher of either 2, 3, or 5mg weekly PO that results in less than a 33% incidence of DLT.

Note: Based on evaluation of the safety and tolerability data gathered during the dose determination

phase together with data from other clinical trials, it may also be decided that accrual will take

place at an alternate dose level or dosing schedule via a protocol amendment.

Up to 18 patients are expected to be enrolled in the Dose Determination Phase of the study.

3.2 Phase 2 Expansion Phase

The phase 2 expansion phase is a randomized, multicenter, double-blind, placebo-controlled study

phase. Randomization for this portion of the study is stratified by geographic location (US vs. rest

of world).

70 eligible patients are randomly assigned in a 1:1 ratio to either:

• Entinostat per os (p.o.) weekly at the RP2D combined with atezolizumab at a fixed

dose of 1200 mg iv every 3 weeks

OR

Placebo combined with atezolizumab at a fixed dose of 1200 mg iv every 3 weeks

Patients will follow the same schedule of study visits and assessments as specified in the Dose

Determination Phase (with the exception of the tumor tissue biopsy at C2D15). Patients may

continue study treatment until documented progressive disease, intolerable toxicity or meets one of the study withdrawal criteria (Protocol Section 11).

Patients will be followed for overall survival (OS) until death (due to any cause) or the Sponsor terminates the trial.

#### 4. STUDY ENDPOINTS

#### 4.1 Phase 1b Dose Determination Phase

The primary endpoint of the Phase 1b Dose Determination portion of the study is the determination of the DLT, MTD or RP2D of entinostat in combination with atezolizumab at the dose of 1200mg. The following safety endpoints will also be assessed:

- AEs
- Clinical laboratory parameters, vital signs, physical examinations, and ECGs

Exploratory endpoints will also be assessed and are discussed in a separate SAP.

### 4.2 Phase 2 Expansion Phase

#### 4.2.1 Primary Efficacy Endpoint

The primary efficacy endpoint is PFS as determined by the local investigator using RECIST 1.1.

# 4.2.2 Secondary Efficacy Endpoints

- PFS determined by the local investigator using irRECIST
- ORR (CR or PR) by RECIST 1.1
- ORR (irCR or irPR) by irRECIST
- CBR (CR, PR or SD for at least 24 weeks) by RECIST 1.1
- CBR (irCR, irPR, or irSD for at least 24 weeks) by irRECIST
- OS

In patients who experience a response to treatment based on RECIST 1.1 (CR or PR) or on irRECIST (irCR or irPR):

- DOR
- TTR

4.2.3 Safety

Safety endpoints are:

• AEs

Clinical laboratory parameters, vital signs, physical examinations, and ECGs

4.2.4 Exploratory

The exploratory endpoints will be discussed in separate SAP(s).

5. STATISTICAL CONSIDERATIONS

5.1 Hypothesis for Phase 2

The primary efficacy analysis will be the comparison of the distribution of PFS between the two treatment groups using a stratified logrank test at one-sided 10 % level of significance, i.e.:

 $H_0$ : PFS in experimental arm (entinostat + atezolizumab) = PFS in control arm (placebo + atezolizumab)

VS.

H<sub>a</sub>: PFS in experimental arm (entinostat + atezolizumab) > PFS in control arm (placebo + atezolizumab)

5.2 Sample Size

5.2.1 Phase 1b Dose Determination Phase

Three to six patients will be enrolled in each dose cohort based on a standard Phase 1 dose-finding scheme.

A starting sample size of 3 evaluable patients per dose cohort, expanding to 6 in the event of a marginal DLT rate (33%) was deemed to be a safe and conventional approach in dose-finding. Assuming a true DLT rate of 5% or less, there would be a 3% chance that dose escalation would be halted in a given cohort (i.e. observing 2 or more patients with DLT). If a true DLT rate of 50% is assumed, then there would be an 83% chance that dose escalation would be halted in a given cohort.

6 patients will need to be treated in a dose level for it to be considered as MTD or RP2D.

Patients who discontinued the study for reasons other than study drug related toxicities before

completing Cycle 1 will be replaced.

Therefore, between 6 and 18 patients will be included in the Dose Determination Phase.

5.2.2 Phase 2 Expansion Phase

The following assumptions are made:

• Patients in the control arm have true median PFS of 4 months

• Patients in the experimental arm have true median PFS of 7 months (under exponential

distribution, true PFS hazard ratio of 0.57)

• Expected accrual duration will be 9 months and an additional 9 months of follow-upThe α

type I error rate is set to 10% (1-sided)

• The  $\beta$  type II error rate is set to 20% (i.e. the power of the trial will be 80%)

Under these assumptions, 70 patients (35 per arm) will be enrolled in the trial, which is projected to

result in 60 PFS failures, defined as documented disease progression by RECIST 1.1 or death due

to any cause without documented disease progression beforehand, within approximately 18 months

of the first patient randomized.

It is anticipated that the number of patients that drop out without PFS failure will be low (2-3%).

Depending on the actual number of such dropouts, the number of patients accrued maybe increased

by 6-10 patients to accommodate for a higher-than-expected number of dropouts.

5.3 Randomization and Stratification

The randomization technique used for the study is a stochastic minimization, using

minimization probability parameter of 0.80. The randomization is performed via ID-net

(which is the IWRS from IDDI).

Prior to dosing, eligible patients are randomized in a 1:1 ratio into 2 treatment arms,

stratified by geographic location.

5.4 Timing of Analyses

5.4.1 Phase 1b Dose Determination Phase

A safety analysis will be performed at the completion of the dose determination phase.

Document owner(s): Document ID: DM-025-037 Version: 1.0 – Final – 08-Jun-2017 

5.4.2 Phase 2 Expansion Phase

The following analyses are planned:

• An interim safety analysis will be performed following the completion of Cycle 1 for the

first 20 patients enrolled in the Phase 2 expansion phase, and will utilize a Data Safety

Monitoring Board (DSMB).

An interim efficacy analysis will be performed when 45 PFS events have observed. Data

cut-off for the analysis will be based on the calendar date of the 45th PFS event (per

RECSIT 1.1). Safety and secondary endpoints will also be evaluated. The same data cut-off

used for the PFS analysis is also used for the corresponding analysis of safety and

secondary endpoints.

• Primary efficacy analysis will be performed when 60 PFS events are observed. Similarly,

the data cut-off for the primary analysis will be based on the calendar date of the 60th PFS

event. Safety and secondary endpoints will coincide with the primary PFS analysis.

• End of study analysis for safety and OS analysis will be performed when the last patient

terminates study treatment.

6. **DEFINITIONS** 

6.1 Progression-Free Survival (PFS)

The duration of PFS, defined as the number of months from randomization to the earlier of

progressive disease or death due to any cause. One month is considered 30.4375 days.

PFS (months) = (Date of Progression or Censoring – Date of Randomization + 1) ÷ 30.4375

Patients who meet one or more of the following conditions at the time of primary analysis will be

censored:

No screening or post-screening disease assessments unless death occurred prior to the first

planned assessment.

• Initiation of a new anticancer therapy in the absence of documented progression.

• Death or progressive disease after missing 2 or more consecutively scheduled disease

assessment visits

• Last known to be alive and progression-free on or before the data cut-off date

The following table, adopted from FDA guidance "Guidance for Industry Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics" (May 2007) illustrates how the cases will be handled for primary analysis. If a patient is censored satisfying more than one criteria, the situation with the earliest date will be considered.

Table 1 – Primary Rules for Determining Date of Progression or Censor for Primary Progression-Free Survival

| | Situation | Date of Progression or | Outcome |
|---|---|---|---|
| | | Censoring | |
| 1 | Death before first PD assessment | Date of death | Progressed |
| 2 | Death or disease progression<br>between planned disease<br>assessments | Date of death or first disease assessment showing disease progression, whichever occurs first | Progressed |
| 3 | No baseline tumor assessments | Date of randomization | Censored |
| 4 | New anticancer treatment started (in absence of documented progression) | Date of last radiological assessment of measured lesions prior to the start of the new anticancer treatment | Censored |
| 5 | Death or progression after more than 2 or more consecutive visits | Date of last radiological assessment of measured lesions without documented disease progression that is before the first missed visit | Censored |
| 6 | Last known to be alive and progression-free on or before the data cut-off date | Date of last radiological assessment of measured lesions | Censored |

The following sensitivity analyses will also be provided:

Table 2 - Progression-Free Survival Sensitivity Analysis

| Analysis # | Definition and/or changes from primary analysis; unless otherwise stated, the same PFS censoring rules will be applied |
|---|---|
| 1 | Per-protocol analysis set, instead of full analysis set |
| 2 | PFS events occurring immediately after two or more missing visits will not be censored |
| 3 | Patients who discontinue treatment due to any reason other than disease progression or death are censored at the date of last tumor assessment prior to (or at) treatment discontinuation |
| 4 | Patients who received new anticancer treatment without documented progression will not be censored |
| 5 | Worst case analysis: A patient who is lost to follow-up (or withdrew consent from study participation) before documented progression will be considered progressed at first scheduled radiological assessment date after lost to follow-up (or withdrew consent) (i.e. last radiological assessment + 42 days) |

All analyses described above will use the same methodologies as the primary analysis, except changes as noted in the second column. Each analysis will modify only the rule as stated in the specific row; i.e. rows will not be combined unless otherwise specified.

# 6.2 Objective Response Rate (ORR)

ORR is defined as the crude proportion of patients achieving a best overall response of CR or PR assessed using RECIST 1.1. The best overall response assessed using irRECIST will also be analyzed separately and the corresponding ORR will be calculated. The overall response will be determined locally by the investigator at each scheduled assessment.

Per protocol (Section 10.3.1.3), partial or complete response should be confirmed by a repeat tumor imaging assessment not less than 4 weeks from the date the response was first documented.

The following table will be followed to assign a <u>best</u> overall response based on the achievement and confirmation of two consecutive assessments according to RECIST 1.1:

| Overall response<br>First time point | Overall response Subsequent<br>time point<br>(at Least 4 Weeks Later) | Best Overall Response |
|---|---|---|
| CR | CR | CR |

| Overall response<br>First time point | Overall response Subsequent<br>time point<br>(at Least 4 Weeks Later) | Best Overall Response |
|---|---|---|
| CR | PR | PR |
| CR | SD | SD |
| CR | PD | PD |
| CR | NE | SD |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | PD |
| PR | NE | SD |

$$ORR_{RECIST1.1} = \frac{\# of \ patients \ with \ best \ overall \ response \ as \ CR \ or \ PR}{Total \ number \ of \ patients}$$

Similarly, irCR or irPR based on irRECIST will also be confirmed.

The following table is therefore used for best overall response based on irRECIST:

| Overall response<br>First time point | Overall response Subsequent<br>time point<br>(at Least 4 Weeks Later) | Best Overall Response |
|---|---|---|
| irCR | irCR | irCR |
| irCR | irPR | irPR |
| irCR | irSD | irSD |
| irCR | irPD | irPD |
| irCR | irNE | irSD |
| irPR | irCR | irPR |
| irPR | irPR | irPR |
| irPR | irSD | irSD |
| irPR | irPD | irPD |
| irPR | irNE | irSD |

And ORR based on irRECIST is calculated as follows:

$$ORR_{irRECIST} = \frac{\# of \ patients \ with \ best \ overall \ response \ as \ irCR \ or \ irPR}{Total \ number \ of \ patients}$$

### 6.3 Clinical Benefit Rate (CBR)

CBR is estimated based on the crude proportion of patients in each treatment arm whose best overall response during the course of study treatment is CR, PR or SD lasting for at least 24 weeks (measured from the date of randomization to the last date where SD is reported).

$$CBR_{RECIST\ 1.1} = \frac{\#\ of\ patients\ with\ best\ confirmed\ overall\ response\ as\ CR/PR/\ SD_{lasting\ for > 24\ weeks}}{Total\ number\ of\ patients}$$

Similarly, CBR is calculated based on irRECIST as below:

$$CBR_{irRECIST} = \frac{\# \ of \ patients \ with \ best \ confirmed \ overall \ response \ as \ irCR/irPR/irSD_{lasting.for > 24.weeks}}{Total \ number \ of \ patients}$$

#### 6.4 Overall Survival (OS)

OS is defined as the number of months from randomization to date of death from any cause. Patients who are alive or lost to follow-up as of a data analysis cutoff date will be right-censored. OS (months) = (Date of Death/Censoring – Date of Randomization + 1)  $\div$  30.4375

#### 6.5 Duration of Response (DOR)

DOR is defined as the number of months from the date where a CR / PR (based on RECIST 1.1) or irCR / irPR (based on irRECIST) was firstly observed, to the first date that recurrent or progressive disease is documented. DOR will be calculated for patients who achieved a confirmed CR / PR or irCR / irPR. The same censoring rules for primary analysis will also apply here for patients who achieved a confirmed CR / PR or irCR / irPR. Patients with no baseline or post-baseline assessments will not be analyzed.

```
DOR_{RECIST\ 1.1} (months) = (Date of Progressive Disease – Date of CR/PR + 1) \div 30.4375 DOR_{irRECIST} (months) = (Date of Progressive Disease – Date of irCR/irPR + 1) \div 30.4375
```

#### 6.6 Time to Response (TTR)

TTR is defined for the subset of patients that achieve best overall response of confirmed CR/PR or confirmed irCR/irPR as the number of months from date of randomization to date of the initial documented response of CR/PR (based on RECIST 1.1) or irCR/irPR (based on irRECIST).

Document iD: DM-025-037 Version: 1.0 – Final – 08-Jun-2017

 $TTR_{RECIST 1.1}$  (months) = (Date of CR/PR – Date of Randomization + 1) ÷ 30.4375

TTR  $_{irRECIST}$  (months) = (Date of irCR/irPR – Date of Randomization + 1) ÷ 30.4375

#### 6.7 **Dose-limiting Toxicity (DLT)**

DLT is defined as the occurrence of specific events defined in Section 9.6 of the protocol within the first cycle of treatment (i.e. between Day 1 to Day 21 of Cycle 1) of entinostat in combination with atezolizumab that are considered by the investigator to be at least possibly related to study drug using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

#### 6.8 **Maximum Tolerated Dose (MTD)**

MTD is defined as the highest dose level at which < 33% of 6 patients experience DLT.

#### 6.9 Recommended Phase 2 Dose (RP2D)

RP2D will be equal to or less than the preliminary MTD. This will be determined in discussion with the sponsor, the study medical monitor and dose determination phase investigators.

#### 6.10 Treatment Emergent Adverse Events (TEAEs)

TEAEs is defined as AEs that start on or after the first administration of study treatment or AEs that start before the first administration of study treatment but worsened after study treatment is initiated.

#### **6.11 Other Definitions**

#### 6.11.1 Baseline

The last available assessment done on or before the date of first dose of study treatment.

If patients have no value as defined above, the baseline value will be missing.

### 6.11.2 Date of First Dose

The date of first dose (of study drug) is derived as the first date when a nonzero and nonmissing dose of study drug is administered. This can also be referred to as the start of the study treatment.

#### 6.11.3 Date of Last Dose

The date of last dose (of study drug) is derived as the last date when a nonzero and nonmissing dose of study drug is administered.

#### 6.11.4 Last Contact Date

The last contact date will be derived for patients not known to have died at the analysis cut-off using the latest complete date among the following dates which precede the cut-off date:

- All assessment dates (e.g. vital signs assessment, performance status assessment, tumor assessments, etc.)
- Date patient was last known alive
- Start and stop dates of concomitant medications
- Start and stop dates of adverse events
- Date of last dose
- Date of registration (Phase 1b)/randomization (Phase 2)

#### 7. STUDY POPULATION

# 7.1 Full Analysis Set (FAS)

The Full Analysis Set (FAS) includes all patients who were enrolled (for Phase 1b) or randomized (for Phase 2) to study treatment, regardless of whether they actually received study medication. All efficacy analyses will be evaluated based on data from this population set according to the treatment group they were assigned to at registration/randomization and based on the strata they were originally assigned to at the time of randomization. This population set will be identified using the FASFL (Full Analysis Set Population Flag) as defined in Subject-Level Analysis Dataset (ADSL) according to Analysis Data Model (ADaM).

#### 7.2 Per-protocol Analysis Set

The **Per-protocol Analysis Set** consists of all patients who were enrolled/randomized and did not have any important deviations (i.e. excludes patients with important deviations from FAS). The list of patients who are identified with important deviations will be provided to biostatistician(s) by TRIO Project Management. This population set will be identified using the PPROTFL (Per-Protocol Population Flag) as defined in ADSL according to ADaM.

# 7.3 Safety Analysis Set

The **Safety Analysis Set** consists of all patients who receive any study treatment, and will be used for the analysis of safety data in both Phase 1b and Phase 2 portions of the study. This population will be based on the first dose received at cycle 1, if this differs from that to which the subject was randomized and will be used for the analysis of safety data. This population set will be identified using the SAFFL (Safety Population Flag) as defined in ADSL according to ADaM.

# 8. INTERIM ANALYSIS AND EARLY STOPPING RULE

One interim safety analysis is planned during the Phase 2 of the study after the first 20 patients are treated for one cycle. As mentioned in section 5.3.2, the result of this analysis will be reviewed by DSMB who will act in an advisory capacity to the Sponsor with respect to safeguarding the interests of trial patients and assessing the safety of the interventions administered during the trial. As per Section 13.2 of the protocol, an interim efficacy analysis is performed when 45 PFS events are observed to support the Sponsor's product development plans and ongoing resourcing activities. Although there are no plans to terminate the study early, the DSMB will review the results and decision will be made in collaboration with the Sponsor as well as the Steering Committee should the study needs to be terminated.

# 9. DATA SCREENING AND ACCEPTANCE

## 9.1 General Principles

For the planned analyses, data acceptance will be based on the creation and review of the tables, listings, and figures (TLF) in collaboration with Data Management and Project Management according to TRIO Standard Guideline SG8.1 "Validation of Statistical Analysis". In general, TLF programs will be created prior to a database snapshot or database lock. Dry run(s) of TLF programs will be done in order to review for extreme, unusual, and missing values. Such cases will be identified to Data Management and Project Management for further investigation and potential resolution prior to a snapshot or lock of the database. As data issues are detected, additional procedures might be needed in order to ensure resolution in subsequent data transfer(s).

For the final analysis, all procedures will be run to ensure previously identified data issues have been resolved. The TLF programs will also be run and the outputs will be reviewed to ensure no further data issues are found.

9.2 **Unblinding Plan** 

For the Phase 2 Expansion Phase of this study, all TRIO personnel will be blinded. At the time of

statistical analysis, only the Independent Statistician, who does not work on the study directly, will

be unblinded. He/she will obtain the unblinded randomization file as well as unblinded medication

list in order to unblind the data and perform the analysis accordingly. All relevant unblinded files

will be stored separately on the network and access to the unblinded data will be restricted to the

Independent Statistician only. Refer to TRIO Standard Operating Procedure SOP 5.7 "Blinding and

Unblinding".

9.3 **Data Handling and Electronic Data Transfer** 

All clinical data will be entered directly by the designated users at the site into the database using

Oracle Clinical Remote Data Capture (OCRDC) according to electronic Case Report Form (eCRF)

and will be extracted in the form of raw SAS® datasets by Data Management. Data extracts will be

provided to biostatistician(s) on a regular basis. Once the final data queries have been generated and

resolved, the database will be deemed "locked" and final database extract will be performed after

official data snapshots are completed. The data used for all the analyses will be archived.

9.4 Handling of Incomplete and Missing Data

Missing and incomplete data will be identified for investigation, and possible resolution, by Data

Management and Project Management prior to an official database snapshot or database lock

through review of TLF.

Missing Data: All analyses and descriptive summaries will be based on the reported data. Unless

otherwise specified, missing data will not be imputed or "carried forward."

**Partial or Missing Date for Adverse Events and Concomitant Medications:** 

<u>Imputation Rules for Partial or Missing Stop Dates:</u>

If the month and year are present, impute the last day of that month.

If only the year is present, impute December 31 of that year.

If the stop date is entirely missing, assume the event or medication is ongoing.

If a partial or complete stop date is present and the 'ongoing' box is checked, then it will be

assumed that the adverse event or concomitant medication stopped and the stop date will be

imputed if partial.

## Imputation Rules for Partial or Missing Start Dates

| | | | | Stop Date | | | | |
|---|---|---|---|---|---|---|---|---|
| Complete: yyyymmdd | | Partial: yyyymm | | Partial: yyyy | | Missing | | |
| Start Date | ı | <1st<br>dose | ≥1 <sup>st</sup> dose | < 1 <sup>st</sup> dose yyyymm | $\geq 1^{\rm st}$ dose $yyyymm$ | < 1 <sup>st</sup> dose | $\geq 1^{st}$ dose $yyyy$ | |
| Partial: | = 1 <sup>st</sup> dose yyyymm | 2 | 1 | 2 | 1 | n/a | 1 | 1 |
| уууутт | ≠ 1 <sup>st</sup> dose yyyymm | | 2 | _ | 2 | 2 | 2 | 2 |
| Partial: | = 1 <sup>st</sup> dose | 3 | 1 | 3 | 1 | n/a | 1 | 1 |
| уууу | ≠ 1 <sup>st</sup> dose yyyy | | 3 | | 3 | 3 | 3 | 3 |
| Missing | | 4 | 1 | 4 | 1 | 4 | 1 | 1 |

- 1 = Impute the date of first dose
- 2 = Impute the first of the month
- 3 = Impute January 1 of the year
- 4 = Impute January 1 of the stop year

#### 9.5 Outliers

Outliers will be identified through a review of TLF for investigation by Data Management and Project Management. All outlier data will be included in the analyses presented in this SAP. Any unconfirmed outlier data will be followed up by Project Management.

#### 9.6 Validation Plan

SAS® version 9.3 on the Windows system will be used for all TLF creation. The verification of the outputs, the analysis datasets as well as the review of all programs and macros created specifically for this study, will be conducted as outlined in TRIO Standard Operating Procedures SOP 8.3 "Conduct of Statistical Analysis", SOP 8.4 "Preparation of Statistical Analysis" and Standard Guidelines SG 8.1 "Validation of Statistical Analysis".

#### 10. STATISTICAL METHODS OF ANALYSIS

Categorical variables will be summarized in frequency tables, with the counts and percentage of patients in each category. Percentages given in the summary tables will be rounded and thus may not always add up to exactly 100 percent. For continuous variables, summary statistics will include number of patients, mean, standard deviation, first quartile (Q1), median, third quartile (Q3), minimum and maximum values (range).

# 10.1 Patient Disposition

The patient disposition will be tabulated using the FAS. Frequency count and respective percentages of patients who were in each analysis set (i.e. FAS, Per-protocol, and Safety), and discontinued from treatment and/or study will be summarized by treatment group. The reason for discontinuation (from treatment and/or from study participation where applicable) will be summarized considering the categories specified in the case report forms. Listings of disposition information and analysis population will be provided as well.

Protocol Deviation including eligibility deviations of the inclusion/exclusion criteria will be summarized and listed for FAS, by treatment group.

The stratifications factor (for Phase 2 portion) will also be tabulated by treatment group.

#### 10.2 Demographics and Disease Characteristics

The following demographics and baseline characteristics will be summarized and listed for the FAS by treatment group:

### **Demographics:**

- Age, INT (Date of enrollment/randomization Date of birth) / 365.25)
  - $\circ$  *INT* = *integer part*
  - o Since only the year of birth is collected (YYYY), we assume the full date to be 31-Dec-YYYY
- Race
- Ethnicity
- Menopausal Status
- Weight at Baseline
- Height at Baseline
- ECOG Status at Baseline

#### **Disease Characteristics:**

• Time from Initial Diagnosis to Randomization

• Primary Tumor Location

• Staging at Initial Diagnosis

• Histopathological Type at Initial Diagnosis

Histopathological Grade at Initial Diagnosis

• Disease Status at Registration

• Time from Metastatic / Locally Recurrent Disease to Randomization

• Local Estrogen Receptor Status

Local Progesterone Receptor Status

• Local HER2 Status

10.3 Prior Surgery for Breast Cancer

Number of patients who underwent prior surgeries will be summarized by type and location of surgery. A listing will also be provided.

10.4 Prior Systemic Anti-Cancer Therapy

Number of regimens of prior systemic anti-cancer therapies will be summarized by type and indication. A listing will be provided to show the specifics of the therapies.

10.5 Prior Radiation Therapy

Number of radiation therapies will be summarized by site and indication. A listing will be provided to show the specifics of all reported radiation therapies.

10.6 Medical History

The medical history is coded by the most current version of Medical Dictionary for Regulatory Activities (MedDRA), and will be summarized for FAS by System Organ Class (SOC) and Preferred Term (PT) by treatment group.

10.7 Extent of Exposure

Number of Cycles, Duration of Treatment, Cumulative Dose and Relative Dose Intensity (RDI) will be summarized by treatment for the safety analysis set.

Atezolizumab:

- Number of Cycles: number of cycles having total dose > 0 mg reported
- Duration of Treatment (weeks) =  $[(Date of last dose date of first dose) + 21] \div 7$
- Cumulative Dose (mg) = sum of total dose administered as reported
- Weekly Dose Intensity (mg/week) = (Cumulative Dose) ÷ (Duration of Treatment)
- Planned Weekly Dose Intensity (mg/week) = 1200mg ÷ 3 weeks = 400
- RDI (%) = (Weekly Dose Intensity ÷ Planned Weekly Dose Intensity) × 100

#### **Entinostat:**

- Number of Cycles: number of cycles having total dose > 0 mg reported
- Duration of Treatment (weeks) =  $[(Date of last dose date of first dose) + 21] \div 7$
- Cumulative Dose (mg) = sum of total dose administered as reported
- Weekly Dose Intensity (mg/week) = (Cumulative Dose) ÷ (Duration of Treatment)
- Planned Weekly Dose Intensity (mg/week) = (Dose Cohort as assigned in Phase 1b or RP2D in Phase 2) ÷ 3 weeks
- RDI (%) = (Weekly Dose Intensity ÷ Planned Weekly Dose Intensity) × 100

The RDI will be additionally presented categorized (i.e., number and percentage of patients with RDI of < 60%, 60 - < 80%, 80 - < 90%, 90 - < 110%, > 110%).

The number and percentage of patients with dose interruptions/discontinuations or reduced (entinostat/placebo at Phase 2 only), along with their respective reasons will be summarized.

For entinostat/placebo, the compliance will be summarized by visit using the following calculation:

$$Compliance~(\%) = \frac{\textit{Number of Tabs taken} + \textit{Number of Tabs Returned}}{\textit{Number of Tabs Dispensed}} \times 100$$

## 10.8 Efficacy Analyses

Efficacy data for the primary endpoint and the secondary endpoints will be analyzed for the FAS and, where appropriate, the Per-protocol Set. Sensitivity analyses and subgroup analyses will be conducted as appropriate; refer to Table 2 and Table 3. Summaries and figures of the efficacy endpoints will be generated by treatment group as per randomization.

#### 10.8.1 PFS

The duration of PFS will be summarized descriptively using Kaplan-Meier (KM) curves. Inferential comparisons between treatment arms will be made using stratified log-rank test, stratifying on

Document owner(s):


Document ID: DM-025-037 Version: 1.0 – Final – 08-Jun-2017

Document Location: R:\TRIO025\TMF\G Stats\G01 SAP\DM-025-037 - Statistical Analysis Plan - v1 0 Final - 08-Jun-2017.docx

geographic location (US vs. Rest of World). The KM estimate of the PFS survival distribution function will be computed for each treatment group using PROC LIFETEST with method=KM option in SAS. For each treatment group, the KM estimates for the median PFS time, the first and third quartiles will be presented, along with approximate 95% confidence intervals (CI) calculated using Greenwood's formula. Example of PROC LIFETEST code with and without stratification is presented below:

```
* Unstratified;
proc lifetest data=<PFS> method=km;
  time <pfsmonth>*<pfscens>(1);
  strata <trt>;
run;

* Stratified;
proc lifetest data=<PFS> method=km;
  time <pfsmonth>*<pfscens>(1);
  strata <geographical region> / group= <trt>;
run;
```

The effect of treatment on PFS will also be compared using a stratified Cox proportional hazards model. The hazard ratio with two-sided 95% CI will be derived from the stratified Cox proportional hazards model using PROC PHREG with ties=EXACT option in the model. Homogeneity in the hazard ratios between randomization strata will be examined by Wald's test. The corresponding results without stratification will be reported as supplemental analyses.

Example of PROC PHREG code with and without stratification is presented below:

```
* Unstratified;
proc phreg data=PFS;
class trt(ref='1');
model dfsmonth*dfscens(1)=trt / risklimits ties=exact;
run;

* Stratified;
proc phreg data=PFS;
class trt(ref='1');
model dfsmonth*dfscens(1)=trt / risklimits ties=exact;
strata <geographical region>;
run;
```

Testing of Proportional Hazard assumption will also be done using the following stratified model:

```
proc phreg data=pfs;
  model <pfsmonths>*<pfscens>(1) = <trt> / risklimits Ties=exact;
      assess var=(<trt>) ph / crpanel resample seed=199;
      strata <geographical region>;
  run:
```

Document owner(s):


Document ID: DM-025-037 Version: 1.0 – Final – 08-Jun-2017

In addition, Hazard Ratio for treatment effect will be estimated using a multivariate Cox proportional hazards model to be constructed by selecting variables among all the potential variables listed in the subgroup analysis (see Section 10.10) using stepwise selection method with entry p-value 0.05 and exit p-value 0.1. The treatment factor will be kept out of the model throughout the covariate selection process and only added into the final model. HR for treatment effect and corresponding 95% confidence interval (CI) will be estimated from the final model. Note that a covariate may be removed from the analysis if the number of patients/events representing one level of that variable is insufficient or data collected on that variable are

A sensitivity analysis will be performed to assess the impact of the different censoring mechanisms and deviations from the planned schedule of disease assessments; refer to Table 2.

10.8.2 ORR

insufficient.

The ORR observed in the treatment groups will be compared adjusting for the stratification variables using the Cochran-Mantel-Haenszel (CMH) test using PROC FREQ in SAS. A 95% CI will be calculated by treatment arm for the true ORR.

Example of PROC FREQ for testing ORR is provided below:

```
proc freq data=<ORR>;
   tables <trt> * <Response> / relrisk cmh;
   weight Count;
run;
```

The best overall response outcome (CR/PR/SD/PD/NE) will be summarized and tabulated for the FAS by treatment group.

10.8.3 CBR

The analysis of CBR will be based on the methods described above for ORR.

10.8.4 OS

The analysis of OS will be based on methods described above for PFS.

10.8.5 DOR and TTR

DOR and TTR will be summarized descriptively for each treatment arm using the KM method. Inferential comparisons between treatment arms for DOR and TTR are not planned.

Document owner(s):


Document ID: DM-025-037 Version: 1.0 – Final – 08-Jun-2017
Document Location: R:\TRIO025\TMF\G\_Stats\G01\_SAP\DM-025-037 - Statistical Analysis Plan - v1 0 Final - 08-Jun-2017.docx

10.8.6 Anticancer therapy after end of study treatment

A summary of number of patients received anticancer therapy after end of study treatment will be

tabulated by the type of therapy according to treatment group.

10.9 Safety Analyses

Safety analyses will be performed on the safety analysis set.

10.9.1 Physical Examinations

The number of patients who had done complete and/or symptom-directed physical examinations at

each visit will be tabulated by treatment group.

10.9.2 Adverse Events

The reported AE term will be coded using the current version of the MedDRA. The severity of AE

will be presented as reported by the investigator based on NCI CTCAE version 4.03.

Incidence of TEAE will be tabulated by SOC, PT for:

All TEAEs

• TEAEs by relationship to study treatment and maximum severity grade

• TEAEs with action of study treatment delayed/interrupted or dose reduced

• TEAEs with action of study treatment discontinued

• Serious Adverse Events (SAE) (not Serious TEAEs)

In the event a patient experiences repeat episodes of the same AE, the event with the highest

severity grade and strongest causal relationship to study treatment will be used for purposes of

incidence tabulations.

All AEs leading to deaths will be summarized (not TEAEs). An AE will be considered as leading to

death if it has a grade 5.

Detailed listings for all AEs will be provided. A flag will be used to identify which AE is

considered as treatment emergent.

For the Phase 1b dose determination phase, the observed DLT rate in each dose cohort will be

calculated by the crude proportion of patients who experienced DLT with a 2-sided 95% exact

binomial CI.

10.9.3 Death

All deaths will be reported in a patient listing, which will include the primary cause of death, and

the number of days between the date of last dose to study drug and death.

10.9.4 Laboratory Values

Hematology and serum blood chemistry will be summarized in descriptive statistics by calculating

the mean, standard deviation, median, and range for the following:

Baseline value

Minimum post baseline value

Maximum post baseline value

Average post baseline value

Last post baseline value

Laboratory values will be assigned toxicity grade when available using NCI CTCAE version 4.03.

Shift tables in laboratory toxicity grades (comparing baseline grade with worst post-baseline grade)

will be analyzed using standard shift tables, presenting number and proportion of patients and their

maximum grade shift.

For laboratory tests without a toxicity grading scale, the shift table will present directional shifts

from baseline to above or below the laboratory standard normal range using the maximum increase

and/or decrease observed throughout the course of treatment/observation.

10.9.5 ECOG Performance Status

Tabulation of ECOG Performance Status results will be done for the following:

Baseline value

Minimum post baseline value

Maximum post baseline value

• Last post baseline value

A shift table will be provided as well from baseline status to the worst status of post-baseline time

points.

### 10.9.6 Vital Signs

Vital sign measurements will be summarized by descriptive statistics in the same manner described for laboratory values.

### 10.9.7 Electrocardiogram (ECG)

ECG results will be tabulated in terms of frequency and percentage of patients according to findings reported by investigators at the assessed time points.

#### 10.9.8 Concomitant Medication

Prior and concomitant medications are coded to the current version of World Health Organization Drug Dictionary (WHODD). The generic term will be tabulated and listed by patient.

# 10.10 Subgroup Analysis

Subgroup analyses will be done for PFS and OS to assess internal consistency of study results and whether there is significant treatment heterogeneity across any of the subgroups. Tests within each subgroup and tests for subgroup-by-treatment-interaction terms will use an unstratified test from an unstratified Cox proportional hazards model. Additionally, these subgroup analyses will also be performed using a stratified test/model.

The following subgroup analyses are planned:

**Table 3 – Planned Subgroup Analyses** 

| Subgroup | Reason |
|---|---|
| Geographical region (US vs. Rest of World) | IWRS stratification factor |
| Prior endocrine therapy | Baseline demographic or prognostic factor |
| Prior chemotherapy | Baseline demographic or prognostic factor |
| Prior adjuvant/neoadjuvant systemic anticancer therapy | Baseline demographic or prognostic factor |
| ECOG 0 vs. ECOG 1 | Baseline demographic or prognostic factor |
| Disease stage at study entry: unresectable locally recurrent vs. metastatic | Baseline demographic or prognostic factor |
| Number of metastatic sites: $\geq 3$ vs. $\leq 3$ (based on the location/organ; i.e. 3 liver lesions count | Baseline demographic or prognostic factor |


| as 1 metastatic site) | |
|---|---|
| Disease-free interval: none, < 24 months, vs. > | |
| 24months (based on the first surgery expected to | Baseline demographic or prognostic factor |
| be curative, to the first relapse/progression date) | |

# 10.11 Pharmacokinetic and Antidrug Antibody Analyses –

It will be done in a separate document.

# 10.12 Correlative Analyses

It will be done in a separate document.

# 11. LIST OF PLANNED TABLES, FIGURES, LISTINGS

# 11.1 Planned Tables

| Title | Population | Description |
|---|---|---|
| Patient Disposition | FAS | Tabulates the disposition of all patients by treatment |
| | | group, including the number of patients in each |
| | | population set as well as the number of patients |
| | | discontinued from study treatment, and the number of |
| | | patients discontinued from study. The reason for drug |
| | | discontinuation and study discontinuation will also be |
| | | summarized. |
| Stratification Factors | FAS | Tabulates the stratification factor (Geographic |
| | | Location – US vs. Rest of World) by treatment group. |
| | | (Phase 2 only.) |
| Protocol Deviations | FAS | Tabulate the number of patients who reported protocol |
| | | deviations by deviation category for each treatment |
| | | group. |
| Eligibility Deviations | FAS | Tabulates the number of patients who violates |
| | | inclusion/exclusion criteria by criterion for each |

| Title | Population | Description |
|---|---|---|
| | | treatment group |
| Baseline Demographics | FAS | Tabulates summary statistics of the demographics (age, race, ethnicity, menopausal status, weight, height and ECOG status at baseline). |
| Disease Characteristics | FAS and Safety | Tabulates summary statistics for time from initial diagnosis to randomization, primary tumor location, staging at initial diagnosis, histopathological type at initial diagnosis, histopathological grade at initial diagnosis, disease status at registration, time from metastatic/locally recurrent disease to randomization, hormonal receptor status, and HER2 status. |
| Prior Surgery for Breast Cancer | FAS | Tabulates the number of patients with type and location of surgery for each treatment group. |
| Prior Systemic Anti-<br>Cancer Therapy | FAS | Tabulates the number of patients by type and indication of the systemic cancer therapy for each treatment group. |
| Prior Radiation Therapy | FAS | Tabulates the number of patients by site and indication of prior radiation therapy for each treatment group. |
| Medical History | FAS | Summarizes medical history by SOC and PT for each treatment group. |
| Study Drug Exposure | Safety | Summarizes the number of cycles, the duration of treatment, cumulative dose, and RDI by treatment group. The number of dose interruptions/discontinuation or reduction will also be summarized. |
| Compliance | Safety | Compliance assessment will be summarized by each visit. |
| Dose Limiting Toxicity | Safety | Tabulates the number of patients experienced DLT |

| Title | Population | Description |
|---|---|---|
| | | and the corresponding DLT at cycle 1 and 2 for each treatment group. For Phase 1b only. |
| Progression-Free<br>Survival | FAS <sup>1</sup> | Summary of PFS results including treatment comparison results. Separate tables will be done for PFS based on RECIST 1.1 and irRECIST. |
| Progression-Free<br>Survival | FAS <sup>1</sup> | Summary of PFS results including treatment comparison results (sensitivity analysis). Separate tables will be done for PFS based on RECIST 1.1 and irRECIST. |
| Objective Response<br>Rate | FAS <sup>1</sup> | Summary of ORR results including treatment comparison results. Separate tables will be done for ORR based on RECIST 1.1 and irRECIST. |
| Clinical Benefit Rate | FAS <sup>1</sup> | Summary of CBR results including treatment comparison results. Separate tables will be done for CBR done based on RECIST 1.1 and irRECIST. |
| Overall Survival | FAS <sup>1</sup> | Summary of OS results by treatment group. |
| Duration of Response ( those with CR/PR or irCR/irPR | FAS <sup>1</sup> | Summary of DOR results by treatment group. |
| Time to Response (same comment as above) | FAS <sup>1</sup> | Summary of TTR results by treatment group. |
| TEAEs Overview | Safety | Tabulates the number of patients with TEAEs, Related TEAEs, Grade 3 / 4 TEAEs, TEAEs with action taken as dose reduced or drug interrupted, TEAEs leading to drug withdrawn, SAE, Fatal AE. For Phase1b, the DLT rate will be presented. |

| Title | Population | Description |
|---|---|---|
| TEAEs | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs | Safety | Summary by PT for each treatment group ordered by |
| | | frequency. |
| TEAEs per Maximum<br>Grade | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs Related to Entinostat | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs Related to<br>Entinostat per<br>Maximum Grade | Safety | Summary by SOC and PT for each treatment group. |
| Grade 3 / 4 TEAEs | Safety | Summary by SOC and PT for each treatment group. |
| Grade 3 / 4 TEAEs | Safety | Summary by PT for each treatment group ordered by |
| | | frequency. |
| TEAEs Related to Atezolizumab | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs Related to<br>Atezolizumab per<br>Maximum Grade | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs Related to<br>Entinostat and/or<br>Atezolizumab | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs Related to<br>Entinostat and/or<br>Atezolizumab per<br>Maximum Grade | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs with Action<br>Taken as Treatment<br>delayed/interrupted for<br>Entinostat | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs with Action<br>Taken as Treatment<br>delayed/interrupted for<br>Atezolizumab | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs with Action<br>Taken as Dose Reduced | Safety | Summary by SOC and PT for each treatment group. (For Phase 2 only) |

| Title | Population | Description |
|---|---|---|
| for Entinostat | | |
| TEAEs Leading to<br>Treatment<br>Discontinuation | Safety | Summary by SOC and PT for each treatment group. |
| TEAEs Leading to<br>Treatment<br>Discontinuation | Safety | Summary by PT for each treatment group ordered by frequency. |
| SAE | Safety | Summary by SOC and PT for each treatment group. |
| AEs Leading to Death | Safety | Summary by SOC and PT for each treatment group. |
| Laboratory Values | Safety | Summary of each laboratory parameter at baseline, minimum post baseline value, maximum post baseline value, average post baseline value and last post baseline value for each treatment group. In addition, shift tables will be presented. |
| ECOG Performance<br>Status | Safety | Summary of ECOG performance status at each baseline, minimum post baseline value, maximum post baseline value, last post baseline value for each treatment group. In addition, a shift table will be presented. |
| Vital Signs | Safety | Summary of descriptive statistics for each vital sign measurements will be done for baseline value, minimum post baseline value, maximum post baseline value, average post baseline value, and last post baseline value for each treatment group. |
| ECG | Safety | Tabulate the frequency and percentage of patients according to findings reported at each time point for each treatment group. |
| Prior and Concomitant<br>Medications | Safety | Tabulate the frequency and percentage of patients according to generic name. Summary will be presented separately for prior medications and |

| Title | Population | Description |
|---|---|---|
| | | concomitant medications. |
| Anticancer Therapy<br>Received after end of<br>study treatment | FAS | Tabulate the frequency and percentage of patients according to type of anticancer therapy received after end of study treatment. |

<sup>&</sup>lt;sup>1</sup> Separate tables to be produced based on per-protocol analysis set if needed.

# 11.2 Planned Listings

| Title | Population | Description |
|---|---|---|
| Screen Failures | N/A | Listing of screen failures and the corresponding reason(s) of failures. |
| Patient Accountability | FAS | Listing of all patients and with population indicators, treatment groups. For patients who discontinued from treatment and/or study, include the reason of respective discontinuations. |
| Demographics | FAS | Listing of demographics. |
| Disease Characteristics | FAS | Listing of disease characteristics. |
| Prior Surgery | FAS | Listing of prior surgery. |
| Prior Systemic Anti-<br>Cancer Therapy | FAS | Listing of prior systemic anti-cancer therapy. |
| Prior Radiation Therapy | FAS | Listing of prior radiation therapy. |
| Study Drug Exposure | Safety | Listing of patients for extent of exposure by visit. |
| Study Drug Exposure<br>Summary | Safety | Listing of patients for summary of exposure (e.g. number of cycles, duration of treatment, cumulative dose, weekly dose intensity, RDI). |
| Efficacy Parameters | FAS | Listing of all efficacy parameters for each patient, including PFS, OS, best overall response, duration of response, and time to response. |
| Tumor Assessment | FAS | Listing of tumor assessment including lesion number, date of assessment, lesion measurement/response, and time-point overall response assessed by RECIST 1.1 and irRECIST. |
| Anticancer Treatment<br>Received after End of<br>Study Treatment | FAS | Listing of anticancer therapies received after end of study treatment; the listing includes the type of therapy, start date, end date (or ongoing) |
| AEs | Safety | Listing of all AE for each patient; the listing includes<br>the verbatim term, PT, SOC, seriousness, worst grade,<br>start date, outcome, stop date, relationship to study<br>drug, action taken for study drug, and treatment |

| Title | Population | Description |
|---|---|---|
| | | emergent flag. |
| TEAEs Related to Entinostat | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| TEAEs Related to<br>Atezolizumab | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| TEAEs Related to Entinostat and/or Atezolizumab | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| TEAEs with Action Taken for Drug Interrupted for Entinostat | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| TEAEs with Action<br>Taken for Dose Reduced<br>for Entinostat | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| TEAEs with Action Taken of Drug Interrupted for Atezolizumab | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| TEAEs Leading to Study<br>Treatment<br>Discontinuation | Safety | Listing of TEAEs in this category using the same structure as the AEs listing with the omission of treatment emergent flag. |
| SAEs | Safety | Listing of TEAEs in this category using the same structure as the AEs listing. |
| AEs Leading to Death | Safety | Listing of TEAEs in this category using the same structure as the AEs listing. |
| Deaths | Safety | Listing of patients who died, including primary cause of death, date of death, date of last dose, and the number of days from date of last dose to death. |
| Laboratory Values | Safety | Listing of all laboratory values and their assigned toxicity grade (where applicable). |
| ECOG Performance<br>Status | Safety | Listing of ECOG at each assessment. |
| Vital Signs | Safety | Listing of all vital signs results at each assessment. |
| Prior and Concomitant<br>Medications | Safety | Listing of all prior and concomitant medications; the listing includes verbatim product name, generic name, start date, end date (or ongoing) and indication. |
| Post Study Follow-up | Safety | Listing of patients who are being followed in post |

| Title | Population | Description |
|-------|------------|-------------------------|
| | | study follow-up visits. |

# 11.3 Planned Figures

| Title | Population | Description |
|-------|------------|----------------------------------------------------|
| PFS | FAS | KM plot of PFS by treatment group. |
| | | Forest plots are done for subgroup analyses. |
| OS | FAS | KM plot and Forest plots of OS by treatment group. |
| DOR | FAS | KM plot of DOR by treatment group. |
| TTR | FAS | Swimmer plot of TTR by treatment group. |
| BOR | FAS | Waterfall plot and Spider plot of BOR for RECIST |
| | | and irRECIST by treatment group. |